CLINICAL TRIAL: NCT01179139
Title: Pathogenesis of Chronic Sinusitis in Relationship to Tobacco Smoke Exposure
Acronym: FAMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Daniel Hamilos MD, M.D., Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2003P002050
Record Dates: First submitted 2010-04-15; First posted 2010-08-11 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Chronic Rhinosinusitis
Keywords: CRS
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Control (Active Comparator)
  Interventions: Other: Biopsy
- CRS (Experimental)
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Percutaneous 2-3 mm biopsies of middle turbinate mucosae and nasal polyps will be obtained with 5 mm Thrucut® (Smith & Nephew, Memphis, TN) biopsy forceps. Generally, 2-3 specimens will be obtained from each side as in previous studies. Healthy controls and subjects with CRS without NP will have biopsies from both middle turbinates. Subjects with CRS with NP will have two nasal polyp biopsies and one middle turbinate biopsy.

SUMMARY:
The purpose of the study is to better understand the causes of chronic rhinosinusitis (CRS)and to determine if being around secondhand cigarette smoke causes swelling in the sinuses. To answer this question, we are inviting healthy volunteers, volunteers with chronic sinusitis, and volunteers with chronic sinusitis with nasal polyposis to complete a questionnaire and undergo a series of tests. These tests will measure their allergies, their exposure to cigarette smoke and the swelling in their sinuses. We are asking you to take part because you are in one of these groups. About 166 people will take part in this research study. All subjects will be enrolled at Massachusetts General Hospital (MGH). The Flight Attendants Medical Research Institute (FAMRI) and the Harvard Clinical and Translational Science Center Harvard Catalyst) are paying for this study.

DETAILED DESCRIPTION:
Chronic sinusitis is one of the most prevalent chronic illnesses in the United States and a significant health concern in terms of public health care expenditure. We wish to learn more about pathogenic factors causing or contributing to chronic sinusitis. One of these factors is secondhand smoke (SS) exposure. However, several other factors are involved, including allergic, environmental, genetic and microbiologic factors and in any given patient, several of these factors may be contributing to the disease. One of our goals is to see whether specific patterns of inflammatory cells, cytokines or chemokines exist that can differentiate these causative factors and to help us to better understand their individual contributions to the disease.

Several inflammatory cells, cytokines and chemokines are present in chronically inflamed sinus tissue, and we believe they form the basis for the disease process. At present, we know very little about what drives them into the sinus tissues. We believe that the types of inflammatory cells, cytokines and chemokines elicited in this disease depend on the inciting stimulus.

Cigarette smoke has well-documented deleterious effects on respiratory mucosa that could promote the development of chronic sinusitis. These include reduction in normal mucociliary function; increased nasal airway resistance; induction of mucin gene expression and induction of chronic inflammation. In the proposed study, we will extend our previous findings to investigate the relationships between SS exposure and these inflammatory markers and also examine the relationship of these cytokines to the expression of particular mucins.

Extracts of cigarette smoke have been shown to induce numerous other proinflammatory effects on respiratory epithelial cells either in vivo or in vitro. In this study we will analyze the gene expression of inflammatory markers in a nasal mucosal biopsy. Our intent is to study sinusitis rather than rhinitis. Nonetheless, we will examine nasal rather than sinus mucosa largely owing to the difficulties posed by obtaining samples directly from the sinuses. Furthermore, recent consensus reports have emphasized the importance of viewing sinusitis as a continuum of nasal and sinus mucosal inflammation. These same arguments have been put forward in terms of the concept of "one airway, one disease" which has emphasized the commonality of mucosal inflammation seen in the upper airway (rhinitis, sinusitis) and the lower airway (asthma). The biopsies will come from the middle turbinate. The latter structure has the same pseudostratified columnar epithelium and a virtually identical appearance to that of maxillary or ethmoid sinus mucosa. We have used biopsies from the middle turbinate in several previous studies of chronic sinusitis, primarily as a comparative tissue representing "healthy" sinus mucosa.

ELIGIBILITY:
Inclusion Criteria:

All of the subjects will satisfy the recently proposed definition for chronic sinusitis, i.e. having symptoms for at least 12 weeks with two or more of the following: anterior and/or posterior mucopurulent drainage, nasal congestion, or facial pain/pressure. Subjects must also have objective evidence of disease on rhinoscopic examination, consisting of (a) thick white or colored mucus from at least one sinus area, (b) edema of the middle meatus or ethmoidal area or (c) the presence of polypoid tissue in the nasal cavity or sinus areas. Sinus CT scans will not be obtained.

Exclusion Criteria:

Subjects with current or past use of cigarettes. Subjects with a history suggestive of immune deficiency (i.e. those who have had > one pneumonia in the past 12 months or those with known immune deficiency) will be excluded. Subjects with a known history of cystic fibrosis, Kartagener's syndrome, immotile cilia syndrome, hypogammaglobulinemia, and individuals taking medications that alter clotting and those with bleeding disorders will also be excluded. Subjects who are pregnant or who have a history of fainting will also be excluded. Subjects who are pregnant, planning to become pregnant, or breastfeeding.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-12; Primary Completion 2010-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Comparison of innate immune and inflammatory factor mRNA expression | 0hr
  To compare the expression profile of innate immune and inflammatory factor mRNA expression in the epithelial and glandular tissue compartments in 8 patients with refractory CRS versus 8 healthy control nasal middle turbinates (HC) using microarray.

SECONDARY OUTCOMES:
Characterization of bacterial microbial community | 0hr
  To characterize and compare the bacterial microbial community in the sinus mucosal tissues from 8 patients with refractory CRS versus 8 HC subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hamilos, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States